CLINICAL TRIAL: NCT06268314
Title: Feeding Pattern and Hypoalbuminemia in Pediatrics With Chronic Kidney Disease.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed Abdel-Gawad, resident doctor, Assiut University
Other Study IDs: hypoalbuminemia in pediatrics.
Record Dates: First submitted 2023-12-25; First posted 2024-02-20 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the impact of feeding pattern on the development of hypoalbuminemia and out come of pediatric patients with chronic kidney disease.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is characterized by an irreversible deterioration of renal function that gradually progresses to end-stage renal disease. During the past 2 decades, the incidence of CKD in children has steadily increased.Children, adolescents, and young adults constitute less than 5% of the end-s population, and their 10-year survival ranges from 70% to 85%.Although children represent only a small proportion of all patients with CKD, affected children pose unique challenges to the health care system and to their providers, who must address not only the primary renal disorder, but the many extrarenal manifestations of CKD that complicate management.Serum albumin is a strong predictor for adverse outcomes in adults with chronic kidney disease (CKD). Because these conditions are amenable to treatments, recognition of hypoalbuminemia and underlying status may improve patient management, potentially leading to better clinical outcomes.Hypoalbuminemia is known to be an independent predictor of survival and hospitalization in adult patients with end-stage renal disease (ESRD) on dialysis.In children with ESRD, a few studies have focused on mortality or hospitalization as outcomes, showing the association of hypoalbuminemia with high mortality in incident dialysis patients and high hospitalization frequency in prevalent dialysis patients.Further, patients with chronic diseases and hypoalbuminemia lose fat-free mass, considered to be an essential indicator of the undernourished state, despite adequate food intake.Protein energy wasting (PEW) is common in patients with CKD and associated with adverse clinical Outcomes .(PEW) is closely associated with malnutrition and inflammation, where serum albumin is an established surrogate biomarker.

Children with CKD are also at high risk of poor nutrition and chronic inflammation .Malnutrition and inflammation are associated with adverse outcomes such as death or hospitalization.Furthermore, among children with CKD, inadequate nutrition is one of the most common causes of growth failure, resulting in short stature or low body mass index (BMI)which is also associated with death or hospitalization.

ELIGIBILITY:
Inclusion Criteria:

The study will include patient on maintenance hemodialysis with hypoalbuminemia according to] Mites SedBuffone GJed Pediatric Clinical Chemistry. 3rd ed., Press(1989)[ (Hypoalbuminemia was defined as an albumin level of less than 3.4 g/dL for patients 7 months or older and less than 2.5 g/dL for patients younger than 7 months. ) who fulfilled the following criteria will be included in the study:

1. Age range from 2-16 years old.
2. Both sexes.
3. On maintenance hemodialysis with hypoalbuminemia

Exclusion Criteria:

1. other causes of hypoalbuminemia such as heart disease, diabetes mellitus , hepatic failure .
2. chronic kidney disease without hypoalbuminemia.

Ages: 2 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Based on determining the main outcome variable ,the estimated minimum required sample size is77. The sample size was calculated using Epi-info version 7 software, based on the following assumptions:
  Main outcome variable is the role of feeding in treating hypoalbuminemia in pediatric patients with CKD . Based on previous studies ( O.S. Catherine. et al. 2002 ) the percentage of patients of chronic kidney disease with hypoalbuminemia53.1% and based on the percentage confidence limits of 7% and a Confidence level =80
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Feeding Pattern and Hypoalbuminemia in Pediatrics With Chronic Kidney Disease. | 2years
  Feeding pattern has important role on improving hypoalbuminemia in pediatrics with chronic renal disease
  Based on determining the main outcome variable ,the estimated minimum required sample size is77. The sample size was calculated using Epi-info version 7 software, based on the following assumptions:
  Main outcome variable is the role of feeding in treating hypoalbuminemia in pediatric patients with CKD . Based on previous studies ( O.S. Catherine. et al. 2002 ) the percentage of patients of chronic kidney disease with hypoalbuminemia53.1% and based on the percentage confidence limits of 7% and a Confidence level =80

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elmenshawy, Study Director — Assist university

REFERENCES:
- [Background] Kalantar-Zadeh K, Cano NJ, Budde K, Chazot C, Kovesdy CP, Mak RH, Mehrotra R, Raj DS, Sehgal AR, Stenvinkel P, Ikizler TA. Diets and enteral supplements for improving outcomes in chronic kidney disease. Nat Rev Nephrol. 2011 May 31;7(7):369-84. doi: 10.1038/nrneph.2011.60. PMID 21629229
- [Background] Palmer SC, Maggo JK, Campbell KL, Craig JC, Johnson DW, Sutanto B, Ruospo M, Tong A, Strippoli GF. Dietary interventions for adults with chronic kidney disease. Cochrane Database Syst Rev. 2017 Apr 23;4(4):CD011998. doi: 10.1002/14651858.CD011998.pub2. PMID 28434208
- [Background] Iseki K, Uehara H, Nishime K, Tokuyama K, Yoshihara K, Kinjo K, Shiohira Y, Fukiyama K. Impact of the initial levels of laboratory variables on survival in chronic dialysis patients. Am J Kidney Dis. 1996 Oct;28(4):541-8. doi: 10.1016/s0272-6386(96)90465-5. PMID 8840944
- [Background] Wong CS, Hingorani S, Gillen DL, Sherrard DJ, Watkins SL, Brandt JR, Ball A, Stehman-Breen CO. Hypoalbuminemia and risk of death in pediatric patients with end-stage renal disease. Kidney Int. 2002 Feb;61(2):630-7. doi: 10.1046/j.1523-1755.2002.00169.x. PMID 11849406
- [Background] Rees L, Mak RH. Nutrition and growth in children with chronic kidney disease. Nat Rev Nephrol. 2011 Sep 27;7(11):615-23. doi: 10.1038/nrneph.2011.137. PMID 21947116
- [Background] Silverstein DM. Inflammation in chronic kidney disease: role in the progression of renal and cardiovascular disease. Pediatr Nephrol. 2009 Aug;24(8):1445-52. doi: 10.1007/s00467-008-1046-0. Epub 2008 Dec 13. PMID 19083024
- [Background] Rees L. 3.21 Nutritional management in children with chronic kidney disease. World Rev Nutr Diet. 2015;113:254-8. doi: 10.1159/000360347. Epub 2015 Apr 13. No abstract available. PMID 25906893